CLINICAL TRIAL: NCT07109622
Title: A Randomized, Double-blind, Placebo-controlled Pilot Study to Evaluate the Efficacy of LN18178 on Improving Sperm Virility (Sperm Motility, Sperm Concentration, and Sperm Morphology)
Brief Title: Effect of Herbal Supplement on Improving Sperm Virility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GENCOR Lifestage Solutions (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: GNC/SV/LN18178/25
Record Dates: First submitted 2025-07-16; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Healthy Human Volunteers
Keywords: Sperm Virility

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LN18178 (Experimental): 400 mg, One capsule to be consumed in the morning after breakfast for 12 weeks.
  Interventions: Dietary Supplement: LN18178
- Placebo (Other): One capsule to be consumed in the morning after breakfast for 12 Weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: LN18178 — 400 mg, One capsule to be consumed in the morning after breakfast for 12 weeks.
  Arms: LN18178
Dietary Supplement: Placebo — One capsule to be consumed in the morning after breakfast for 12 Weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of LN18178 on improving sperm virility.

DETAILED DESCRIPTION:
A total of 40 Males aged between 25-45 years will be included in the study. Assessment of inclusion and exclusion criteria will be done based on clinical and laboratory investigations. The eligible subjects will be randomized as per the computer-generated randomization list. The subjects will be assigned to either LN18178 - 400 mg or placebo arms at 1:1 ratio. The subjects will be instructed to take one capsule daily in the morning after breakfast for 12 weeks. A part from primary and secondary outcomes, the study will also record the vital signs and adverse events to evaluate the herbal composition safety and tolerability. The safety assessment of the LN18178 will also include routine laboratory investigations on blood, urine and clinical chemistry at screening and the final visit of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Males aged between 25-45 years with a Body Mass Index (BMI) of 20-29 kg/m2.
2. Subjects with a history of infertility of at least 12 months despite regular unprotected intercourse.
3. Subjects with semen analysis showing abnormal sperm concentration (< 16 million/ml), progressive motility (< 30%), and total motility (< 42%), normal morphology (< 4%). (WHO guidelines- 6th edition, 2021)
4. Subjects with total testosterone ≥300 ng/dL.
5. Subjects who are willing to abstain from sexual activity that results in ejaculation for 3 to 5 days before semen analysis.
6. Subjects who are in a stable sexual relationship and sexually active during the study.
7. Subjects willing to use contraceptives during study period.
8. Subjects agree to maintain current diet and activity level.
9. No urogenital infection or anatomical abnormality of this system, including varicocele; no prior history of surgery in the pelvic area; no uncontrolled systemic illness, such as liver and gallbladder cancers, renal failure, thyroid disorders, and cerebral haemorrhage; no prior history of trauma to the testes; no unilateral testicular atrophy; no previous history of chemotherapy or treatment with anticoagulants, corticosteroids, testosterone and anti-androgen medications during the 8 weeks before the study.
10. Subject considered generally healthy as per health history and routine clinical investigations during screening.
11. Ability to understand the risks/benefits of the protocol and willing to sign the written informed consent.

Exclusion Criteria:

1. Employees working on night shifts.
2. Subjects with identifiable cause for Oligoasthenoteratozoospermia (OAT) (includes Cryptorchidism, Orchitis and Radiation or chemotherapy etc.).
3. Subjects with Systolic >140 and Diastolic >90 mmHg blood pressure and Fasting blood glucose (FBG) >125 mg/dl.
4. Smokers and alcoholics.
5. Subjects underwent treatment for COVID 19 within the last 3 months or tested positive during the study will be excluded.
6. Subject with any physical disability that may limit sexual function.
7. Subjects with history of taking medications for oligospermia or any other sexual problems, including PDE-5 inhibitors, and dysfunctions related to genito-urinary system, muscular dystrophy and coagulation.
8. Subjects with clinical history of genital surgery, endocrine disorders e.g. hypopituitarism, pituitary tumors, hypo- and hyperthyroidism, hypogonadism, inherited (genetic and chromosomal) disorders, etc.
9. Subjects diagnosed with sleep apnea or related disorders.
10. Subjects consuming medications that can interfere with muscle mass such as corticosteroids, testosterone replacement or anabolic drugs.
11. Subjects who consume recreational drugs (such as cocaine, methamphetamine, marijuana, etc.) or chewable tobacco products.
12. Subjects having history of Benign Prostate Hyperplasia (BPH), stroke, myocardial infarction, coronary artery disease, cardiac failure, angina, life-threatening arrhythmia within the past 6 months.
13. Subjects under medications including vitamins, antidepressants, anticholinergics, inhaled beta agonists, anti- hyperlipidemic, psychotropics etc.
14. Subjects using any centrally acting anorectic agents, drugs that inhibit the absorption of nutrients and endocannabinoid neuromodulators during the two weeks prior to enrolment into the study.
15. Subjects who underwent major surgical procedures in last 6 months, which may affect their quality of life.
16. Subject with HIV positive or any other STDs.
17. History of psychiatric disorder that may impair the ability of subjects to provide written informed consent.
18. Subject has participated in a clinical study within the last 90 days prior to recruitment or concurrently participating in another study.

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males aged between 25-45 years
Enrollment: 40 (Estimated)
Dates: Start 2025-08-08 (Estimated); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Change in motility (% Motile Sperms) using manual microscopic examination. | Screening, weeks 8, 12 & 16
  Assessed through manual microscopic examination according to WHO guidelines. The percentage of motile sperm (progressive + non-progressive) will be calculated. A higher percentage reflects improved reproductive function.

SECONDARY OUTCOMES:
Change in semen Concentration (millions/mL) using manual microscopic examination. | Screening, weeks 8, 12 & 16
  Measured manually using a Makler counting chamber. Concentration is expressed in millions of sperm per milliliter. Higher concentration indicates better fertility potential.
Change from baseline to the end of the study period in Morphology of sperm (% normal forms) using manual microscopic examination. | Screening, weeks 8, 12 & 16
  Assessed through microscopic evaluation following WHO criteria. The percentage of sperm with normal morphology will be reported. Greater % indicates enhanced fertility potential.
Change from baseline to the end of the study period in Sperm DNA fragmentation Index (% DFI) using Sperm Chromatin Dispersion method. | Screening, Weeks 12 & 16
  Assessed using the SCD (Sperm Chromatin Dispersion) method. The DNA Fragmentation Index (DFI) represents the percentage of sperm with fragmented DNA. A decrease in DFI is associated with improved fertilization potential.
Change from baseline to the end of the study period in International Index of Erectile Function (IIEF-15) | Baseline (day 1), Weeks 4, 8,12 & 16
  A validated, self-administered questionnaire consisting of 15 items covering erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction. Each item scored from 0 to 5; total score ranges from 0 to 75. Higher scores indicate better sexual function.
Change from baseline to the end of the study period in Quality of life short form (SF-36) | Baseline (day 1), Weeks 4, 8,12 & 16
  The 36-Item Short Form (SF-36) is a self-reported questionnaire used to assess overall health and quality of life. It consists of 8 domains, each scored on a scale from 0 to 100. Higher scores indicate a better quality of life and improved health status.
Change from baseline to the end of the study period in Serum hormonal biomarkers: Total Testosterone (ng/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  Testosterone is a male sex hormone produced by the gonadal tissue. An increase in both total testosterone levels enhances sexual drive and supports sperm production
Change from baseline to the end of the study period in Serum hormonal biomarkers: Free Testosterone (pg/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  Testosterone is a male sex hormone produced by the gonadal tissue. An increase in both free testosterone levels enhances sexual drive and supports sperm production
Change from baseline to the end of the study period in Serum hormonal biomarkers: Follicle-Stimulating Hormone (mIU/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  Follicle-stimulating hormone (FSH), produced by the pituitary gland, plays a key role in supporting spermatogenesis. Any deviation from normal FSH levels can disrupt sperm production and affect sexual development.
Change from baseline to the end of the study period in Serum hormonal biomarkers: Luteinizing Hormone (mIU/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  Luteinizing hormone (LH), released by the pituitary gland, stimulates testosterone production. Maintenance LH levels within the normal range is important for healthy sexual function.
Change from baseline to the end of the study period in Serum hormonal biomarkers: Inhibin B (pg/ml) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  Inhibin B is produced exclusively by the testes and plays a key role in regulating FSH secretion from the pituitary gland. Improvement in Inhibin B is an indication of healthy testicular volume and an adequate sperm count.
Change from baseline to the end of the study period in Semen oxidative stress markers MDA: Malondialdehyde (ng/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  MDA, an end product of lipid peroxidation. High lipid peroxidation as represented by MDA levels may cause changes in the sperm and diminish fertility. It is reported that the high MDA production in the male with low fertilization rates. Reduction of MDA by using antioxidant therapy was correlated with the improvement of fertilization rates. A decrease high MDA level of semen favours spermatogenesis.
Change from baseline to the end of the study period in Semen inflammation markers IL-6: Interleukin 6 (pg/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  IL-6 is a pro-inflammatory cytokine and high levels of IL-6 in seminal plasma are often linked to decreased sperm motility. Increased IL-6 levels in seminal plasma indicate inflammation in male reproductive tract, that affects sperm quality.
Change from baseline to the end of the study period in Semen oxidative stress markers GSH: Glutathione (µM) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  GSH is a powerful antioxidant that neutralizes harmful free radicals (reactive oxygen species or ROS) within sperm cells. GSH helps maintain the integrity of sperm membranes, including the plasma membrane, which is essential for sperm motility and fertilization. Sperm motility is positively correlated with seminal reduced glutathione (GSH) levels. GSH deficiency has been shown to lead to the instability of the spermatozoa midpiece, thus resulting in defective motility and morphology of the spermatozoa.
Change from baseline to the end of the study period in Semen oxidative stress markers TAC: Total Antioxidant Capacity (mM) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  Low seminal plasma antioxidants have been found to be implicated in reducing sperm concentration, motility and morphology. Total antioxidant capacity (TAC) has shown to be strongly correlated with semen quality and male infertility.
Change from baseline to the end of the study period in Semen inflammation markers TNF-alpha: Tumor Necrosis Factor-Alpha (pg/mL) using Enzyme-Linked Immunosorbent Assay method | Baseline (day 1), Weeks 12 &16
  TNF-alpha, a cytokine involved in inflammation, can negatively impact sperm quality. Studies indicate that elevated TNF-alpha levels in seminal fluid are associated with reduced sperm motility, viability, and increased DNA damage. TNF-alpha can trigger programmed cell death (apoptosis) in sperm cells, leading to a reduction in sperm count.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abbasi B, Molavi N, Tavalaee M, Abbasi H, Nasr-Esfahani MH. Alpha-lipoic acid improves sperm motility in infertile men after varicocelectomy: a triple-blind randomized controlled trial. Reprod Biomed Online. 2020 Dec;41(6):1084-1091. doi: 10.1016/j.rbmo.2020.08.013. Epub 2020 Aug 20. PMID 33032908
- [Background] Shabsigh R, Kaufman JM, Steidle C, Padma-Nathan H. Randomized study of testosterone gel as adjunctive therapy to sildenafil in hypogonadal men with erectile dysfunction who do not respond to sildenafil alone. J Urol. 2004 Aug;172(2):658-63. doi: 10.1097/01.ju.0000132389.97804.d7. PMID 15247755
- [Background] Pandit S, Biswas S, Jana U, De RK, Mukhopadhyay SC, Biswas TK. Clinical evaluation of purified Shilajit on testosterone levels in healthy volunteers. Andrologia. 2016 Jun;48(5):570-5. doi: 10.1111/and.12482. Epub 2015 Sep 22. PMID 26395129
- [Background] Yoon HS, Kim JR, Park GY, Kim JE, Lee DH, Lee KW, Chung JH. Cocoa Flavanol Supplementation Influences Skin Conditions of Photo-Aged Women: A 24-Week Double-Blind, Randomized, Controlled Trial. J Nutr. 2016 Jan;146(1):46-50. doi: 10.3945/jn.115.217711. Epub 2015 Nov 18. PMID 26581682
- [Background] Wang-Polagruto JF, Villablanca AC, Polagruto JA, Lee L, Holt RR, Schrader HR, Ensunsa JL, Steinberg FM, Schmitz HH, Keen CL. Chronic consumption of flavanol-rich cocoa improves endothelial function and decreases vascular cell adhesion molecule in hypercholesterolemic postmenopausal women. J Cardiovasc Pharmacol. 2006;47 Suppl 2:S177-86; discussion S206-9. doi: 10.1097/00005344-200606001-00013. PMID 16794456
- [Background] Forest CP, Padma-Nathan H, Liker HR. Efficacy and safety of pomegranate juice on improvement of erectile dysfunction in male patients with mild to moderate erectile dysfunction: a randomized, placebo-controlled, double-blind, crossover study. Int J Impot Res. 2007 Nov-Dec;19(6):564-7. doi: 10.1038/sj.ijir.3901570. Epub 2007 Jun 14. PMID 17568759
- [Background] Srivastava MK, Singh G, Kodur RR, Yalamanchi A. A Combination of Punica granatum Fruit Rind and Theobroma cacao Seed Extracts Enhances Sexual Function in Aging Males in a Randomized, Double-blind, Placebo-controlled Study. Int J Med Sci. 2025 Jan 1;22(2):383-397. doi: 10.7150/ijms.99958. eCollection 2025. PMID 39781534
- [Background] Pandit SL, Yaligar D, Halemane M, Bhat A. A proprietary blend of standardized Punica granatum fruit rind and Theobroma cocoa seed extracts mitigates aging males' symptoms: A randomized, double-blind, placebo-controlled study. Int J Med Sci. 2022 Jul 11;19(8):1290-1299. doi: 10.7150/ijms.73645. eCollection 2022. PMID 35928723
- [Background] Sreeramaneni PGA, Yalamanchi A, Konda MR, Cherukuri SHV, Maroon JC. A Proprietary Herbal Blend Containing Extracts of Punica granatum Fruit Rind and Theobroma cocoa Seeds Increases Serum Testosterone Level in Healthy Young Males: A Randomized, Double-Blind Placebo-Controlled Study. J Diet Suppl. 2023;20(3):411-427. doi: 10.1080/19390211.2022.2035037. Epub 2022 Feb 6. PMID 35129040
- [Background] Madireddy RK, Alluri KV, Somepalli V, Golakoti T, Sengupta K. Toxicological Assessments of a Proprietary Blend of Punica granatum Fruit Rind and Theobroma cacao Seed Extracts: Acute, Subchronic, and Genetic Toxicity Studies. J Toxicol. 2022 May 6;2022:3903943. doi: 10.1155/2022/3903943. eCollection 2022. PMID 35571381
- [Background] Asiedu-Gyekye IJ, Frimpong-Manso S, N'guessan BB, Abdulai Seidu M, Osei-Prempeh P, Kwaku Boamah D. Macro- and Microelemental Composition and Toxicity of Unsweetened Natural Cocoa Powder in Sprague-Dawley Rats. J Toxicol. 2016;2016:4783829. doi: 10.1155/2016/4783829. Epub 2016 Aug 17. PMID 27610134
- [Background] Boroujeni SN, Malamiri FA, Bossaghzadeh F, Esmaeili A, Moudi E. The most important medicinal plants affecting sperm and testosterone production: a systematic review. JBRA Assist Reprod. 2022 Aug 4;26(3):522-530. doi: 10.5935/1518-0557.20210108. PMID 35234023
- [Background] Krausz C. Male infertility: pathogenesis and clinical diagnosis. Best Pract Res Clin Endocrinol Metab. 2011 Apr;25(2):271-85. doi: 10.1016/j.beem.2010.08.006. PMID 21397198
- [Background] Al Wattar BH, Rimmer MP, Teh JJ, Mackenzie SC, Ammar OF, Croucher C, Anastasiadis E, Gordon P, Pacey A, McEleny K, Sangster P. Pharmacological non-hormonal treatment options for male infertility: a systematic review and network meta-analysis. BMC Urol. 2024 Jul 29;24(1):158. doi: 10.1186/s12894-024-01545-1. PMID 39075435
- [Background] Jo J, Lee SH, Lee JM, Jerng UM. Semen Quality Improvement in a Man with Idiopathic Infertility Treated with Traditional Korean Medicine: A Case Report. Explore (NY). 2015 Jul-Aug;11(4):320-3. doi: 10.1016/j.explore.2015.04.007. Epub 2015 Apr 28. PMID 26025007
- [Background] Terai K, Horie S, Fukuhara S, Miyagawa Y, Kobayashi K, Tsujimura A. Combination therapy with antioxidants improves total motile sperm counts: A Preliminary Study. Reprod Med Biol. 2019 Nov 28;19(1):89-94. doi: 10.1002/rmb2.12308. eCollection 2020 Jan. PMID 31956290